CLINICAL TRIAL: NCT00225238
Title: The Effect of Esomeprazole (Nexium) on the Incidence and Severity of Gastrointestinal Adverse Events Associated With a Colonoscopy Purgative
Brief Title: The Effects of Nexium on the Side Effects Associated With a Colonoscopy Prep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 03C.433
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Nausea; Vomiting; Abdominal Pain
Keywords: colonoscopy prep
MeSH Terms: conditions — Nausea; Vomiting; Abdominal Pain | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: esomeprazole (PPI)

SUMMARY:
The purpose of this study is to ascertain if the use of Nexium for 7 days prior to taking a colon prep for a colonoscopy will decrease the side effects that are associated with the colon preparation

DETAILED DESCRIPTION:
The high incidence for colon cancer make it an ideal target for screening. In the United Staes there are approximately 100,00 new cases of colon cancer yearly. Typically the progression from polyps to cancer requires years. This permits a screening procedure to identify polyps befoere they are cancerous. Colon cleansing is required prior to colonoscopy. The gastrointestinal syptoms associted with colonic preps are common and oftn assoicated wwith upper gastrointestinal disorders including GERD, non-ulcer syspepsia, and gastric dysmotoility such as gastropareesis.

ELIGIBILITY:
Inclusion Criteria:

* Subject 18 or older undergoing out-patient colonoscopy

Exclusion Criteria:

* Pregnant females Use of protein Pump Inhibitor within last 4 weeks Use of prescription strength H-2 Blocker within last 4 weeks Use of over the counter strength H-2 Blocker greater than 2x's a week Hospitalized patients PEG-EL purgative contraindicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Outcome will be measured by use of a symptom survey utilizing an analog scale. This will be done at the screen visit and prior to colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: David Kastenberg, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States